CLINICAL TRIAL: NCT05139784
Title: BeAT1D: Benign Autoimmunity and Type 1 Diabetes
Acronym: BeAT1D
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-61; 2021-A01619-32 (Other: ID RCB)
Record Dates: First submitted 2021-10-29; First posted 2021-12-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Autoimmunity; Lymphocytes; Beta cells; Biomarkers
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stools, lymph nodes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 1 diabetes: As defined by the presence of hyperglycemia and/or islet auto-antibodies.
  Interventions: Other: Biosampling
- Other forms of diabetes or autoimmune endocrinopathy: Type 2 diabetes, ketosis-prone diabetes, familial diabetes, secondary diabetes, immunotherapy-induced diabetes; and/or autoimmune endocrinopathies.
  Interventions: Other: Biosampling
- No diabetes: No diabetes or impaired glucose tolerance; no cancer, infectious or immune pathologies; no other condition related to autoimmune and metabolic alterations that may bias the variables under study.
  Interventions: Other: Biosampling
- Lymphadenectomy planned at the occasion of an abdominal surgery: Patients undergoing a lymphadenectomy during surgery for the treatment of their underlying pathology.
  Interventions: Other: Biosampling

INTERVENTIONS:
Other: Biosampling — Collection of blood and stool specimens; and collection of lymph node specimens for the group undergoing surgical lymphadenectomy.

SUMMARY:
National multi-center non-interventional case-control cohort study with collection of biological samples to characterize the autoimmune T and B lymphocytes involved in the development of type 1 diabetes.

DETAILED DESCRIPTION:
The overall objective of this study is to define the differential characteristics of autoimmune T and B lymphocytes across individuals with T1D, other forms of diabetes or autoimmunity, and no disease. The hypothesis is that the characterization of the autoimmune T and B lymphocytes involved in T1D development may allow us to clarify the pathophysiological mechanisms of disease and to identify novel biomarkers for diagnostic, prognostic and therapeutic follow-up applications.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes: type 1 diabetes, as defined by hyperglycemia and long-term insulin therapy started within 6 months from clinical onset; and/or the presence of at least one anti-islet auto-antibody.
2. Other forms of diabetes or autoimmune endocrinopathy: other forms of diabetes (e.g. type 2, ketosis-prone, familial, secondary, immunotherapy-induced diabetes); and/or other autoimmune endocrinopathies, isolated or multiple.
3. No diabetes: absence of diabetes or impaired glucose tolerance; absence of tumor, infectious or immune pathologies, or other conditions related to autoimmune or metabolic alterations that may bias the variables under study.
4. Lymphadenectomy planned in the frame of an abdominal surgery: pancreatic lymphadenectomy planned at the occasion of an abdominal surgery for the treatment of an underlying condition.

Exclusion Criteria:

For all participants: ongoing pregnancy; known HIV/HCV infection; absence of social security coverage; placement under judicial protection; absence of signature of the informed study consent.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with type 1 diabetes, other forms of diabetes or autoimmune endocrinopathies and participants undergoing surgical lymphadenectomy are recruited among patients referred to participating hospital centers.
  Non-diabetic participants are recruited among patient's family members and via at-large calls for healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To define the frequency and phenotype of autoimmune T lymphocytes reactive to islet antigens in the different study groups. | 6 years
  As measured by flow cytometry and sequencing techniques, with a sample size sufficient to attain a 92% statistical power and 5% alpha risk.
  Frequency will be expressed as number of antigen-reactive T lymphocytes per 100,000 total T lymphocytes (e.g. 20/100,000 or 0.02%).
  Phenotype will be expressed as percent of antigen-reactive T lymphocytes expressing a given phenotype, e.g. 20% naïve (CD45RA+CCR7+).
  These 2 measures will be aggregated by expressing the frequency of antigen-reactive T lymphocytes per 100,000 total T lymphocytes expressing a given phenotype, e.g. 20/100,000 antigen-reactive T lymphocytes with 20% naïve will be expressed as 4/100,000 naive antigen-reactive T lymphocytes.

SECONDARY OUTCOMES:
To define the frequency and phenotype of autoimmune B lymphocytes reactive to islet antigens in the different study groups. | 6 years
  As measured by flow cytometry and sequencing techniques, with a sample size sufficient to attain a 92% statistical power and 5% alpha risk.
  Frequency will be expressed as number of antigen-reactive B lymphocytes per 100,000 total B lymphocytes (e.g. 20/100,000 or 0.02%).
  Phenotype will be expressed as percent of antigen-reactive B lymphocytes expressing a given phenotype, e.g. 20% memory (CD24+CD38-negative).
  These 2 measures will be aggregated by expressing the frequency of antigen-reactive B lymphocytes per 100,000 total B lymphocytes expressing a given phenotype, e.g. 20/100,000 antigen-reactive B lymphocytes with 20% memory will be expressed as 4/100,000 memory antigen-reactive B lymphocytes.
To identify novel islet epitopes recognized by autoimmune T and B lymphocytes. | 6 years
  As measured by a lymphocyte frequency within the expected range, e.g. 1-50/million.
To define the phenotype of these lymphocytes. | 6 years
  As defined by exploratory analyses based on omics techniques.
To define the pathogenicity of these lymphocytes against pancreatic beta cells. | 6 years
  As measured by an in vitro killing of beta-cell targets significantly (e.g. >2-fold) higher than the killing observed with control lymphocytes.
To define the antigen receptors used by these lymphocytes to recognize their target epitopes. | 6 years
  As defined by sequencing techniques and sequence annotation using IMGT and MiXCR. Sequence sharing and similarities across receptors will be measured using MiXCR and stringdist.
To define the correlation between the biomarkers analyzed and insulin secretion. | 6 years
  As measured based on the correlation with fasting C-peptide levels >0.2 nM.
To define the differences between lymphocytes in the blood and those in pancreatic lymph nodes. | 6 years
  As measured using the previous frequency and phenotype readouts.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Mallone, MD PhD, Principal Investigator — INSERM U1016 Cochin Institute
Locations (17):
- France (17):
  - APHP Hôpital Avicenne, Bobigny, Île-de-France Region
  - APHP Hôpital J. Verdier, Bondy, Île-de-France Region
  - APHP Hôpital L. Mourier, Colombes, Île-de-France Region
  - Hôpital Sud Francilien, Corbeil-Essonnes, Île-de-France Region
  - Hôpital Mignot - Service de Pédiatrie, Le Chesnay, Île-de-France Region
  - Hôpital Mignot - Services de Diabétologie/Endocrinologie Adultes, Le Chesnay, Île-de-France Region
  - APHP Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - APHP Hôpital Lariboisière, Paris, Île-de-France Region
  - APHP Hôpital Saint Antoine, Paris, Île-de-France Region
  - APHP Hôpital Pitié-Salpêtrière - Service de Chirurgie, Paris, Île-de-France Region
  - Hôpital Pitié-Salpêtrière - Service de Diabétologie, Paris, Île-de-France Region
  - APHP Hôpital Cochin - Service de Chirurgie, Paris, Île-de-France Region
  - APHP Hôpital Cochin - Service de Diabétologie et Immunologie Clinique, Paris, Île-de-France Region
  - APHP Hôpital Européen G. Pompidou, Paris, Île-de-France Region
  - APHP Hôpital Bichat, Paris, Île-de-France Region
  - APHP Hôpital R. Debré, Paris, Île-de-France Region
  - Hôpital René Dubos, Pontoise, Île-de-France Region